CLINICAL TRIAL: NCT06419413
Title: A Transnational Study to Describe Asthma Patient Clinical Characteristics, Treatment Patterns, Biomarkers and to Identify Phenotypes and Endotypes Associated With Differential Outcomes That May Support Future Development of Personalized Treatment Strategies in Chinese Population
Brief Title: A Translational Study to Describe Clinical Characteristics, Biomarkers and to Identify Phenotypes and Endotypes Associated With Differential Outcomes in Chinese Population
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00186
Record Dates: First submitted 2024-04-25; First posted 2024-05-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Cohort A: approximately 80 healthy participants
- Cohort B: approximately 40 mild asthmatics on as-needed low dose inhaled corticosteroids (ICS)-formoterol, or low dose ICS plus as-needed short-acting β2 agonists (SABA), without the need for other controller medication.
- Cohort C: approximately 160 moderate to severe asthmatics on low or medium dose ICS-long acting β2 agonists (LABA), high dose ICS alone or in combination with LABA .
- Cohort D: approximately 75 asthmatics with protocol defined asthma exacerbation.

SUMMARY:
A Translational Study to Describe Asthma Patient Clinical Characteristics, Treatment Patterns, Biomarkers and to Identify Phenotypes and Endotypes associated with Differential Outcomes that may Support Future Development of Personalised Treatment Strategies in Chinese Population

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years of age
* acceptable FEV1 (according to ATS and ERS)
* compliance with study procedures All Asthma Cohorts
* physician diagnosed Asthma greater or equal to 3 months prior to screening visit

Exclusion Criteria:

* history of alcohol or drug abuse within the past year
* pregnant at time of an assessment
* has an altered mental status at the time of informed consent
* receipt marketed or investigational biologic(s) within 3 months or 5 half-lives prior to visit 1, whichever is longer
* history or current upper or lower respiratory infection or symptoms within 2 weeks of baseline assessments
* terminal diseases and/or organ failure or participants otherwise considered not appropriate for the study participation
* Receipt LTRAs or 5-lipoxygenase (5-LO) inhibitors (eg zileuton and montelukast) within 1 month or 5 half-lives prior to baseline, whichever is longer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of up to 355 participants will be recruited and enrolled into Cohort A (healthy participants), Cohort B (mild asthmatics), Cohort C (moderate to severe asthmatics), and Cohort D (Exacerbation asthmatics). Enrolment will be monitored to, 1) ensure at least 20 current smoker or ex-smoker in Cohort A; 2) ensure at least 40 male participants aged 40 years old or above in Cohort A.
Sampling Method: Non-Probability Sample
Enrollment: 355 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-10-08 (Estimated); Study Completion 2026-10-08 (Estimated)

PRIMARY OUTCOMES:
Descriptive summary of demographic and subject characteristic, clinical characteristics and functional deliverables. | At baseline
  Descriptive summary of demographic and subject characteristic, clinical characteristics and functional deliverables at baseline by study cohorts.
Descriptive summary of biomarker level. | At baseline
  Descriptive summary of biomarker level at baseline by study cohorts.
Statistical clustering of key biomarkers. | At baseline
  Statistical clustering of key biomarkers in moderate to severe asthma cohort.
FEV1 level | At baseline
  Evaluation of lung function via airway limitation
Forced Vital Capacity (FVC) | At baseline
  Evaluation of lung function via airway limitation
Maximal Mid Expiratory Flow (MMEF) | At baseline
  Evaluation of lung function via airway limitation
Airway remodeling | At baseline
  Evaluation of lung structure profile and change
Gas trapping | At baseline
  Evaluation of lung structure profile and change
Computed Tomography (CT) Scan | At baseline
  Evaluation of lung structure profile and change

SECONDARY OUTCOMES:
Mean difference in the biomarker level. | At baseline
  Mean difference in the biomarker level between study cohorts
Statistical association between the biomarker and clinical disease outcomes. | From 2023-2025
  Statistical association between the biomarker and clinical disease outcomes in each asthma cohort.
Mean difference in the biomarker level between different tissues | From 2023-2025
  Mean difference in the biomarker level between different tissues in each asthma cohort.

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - Research Site, Chengdu, Sichuan
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Dongguan
  - Research Site, Foshan
  - Research Site, Guangzhou
  - Research Site, Hainan
  - Research Site, Hohhot
  - Research Site, Huizhou
  - Research Site, Kunming
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Taiyuan
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xuzhou
  - Research Site, Zhanjiang
  - Research Site, Zhaoqing

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/